CLINICAL TRIAL: NCT06042205
Title: ALPHA: A Pilot Study to Evaluate the Initial Safety and Performance of the TISSIUM™ Atraumatic Hernia Repair System (TAHRS) for Laparoscopic Hernia Repair
Brief Title: TISSIUM™ Atraumatic Hernia Repair System (TAHRS) Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tissium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF00006-CLPR-002
Record Dates: First submitted 2023-09-08; First posted 2023-09-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hernia repair (Experimental): There is no comparator for this study. All patients are in the treatment allocated group for hernia repair with TISSIUM™ Atraumatic Hernia Repair System (TAHRS)
  Interventions: Device: TISSIUM™ Atraumatic Hernia Repair System (TAHRS)

INTERVENTIONS:
Device: TISSIUM™ Atraumatic Hernia Repair System (TAHRS) — The TAHRS is intended for fixation of prosthetic material to soft tissue

SUMMARY:
The purpose of this study is to capture preliminary clinical safety and performance on the TAHRS

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is 18 years old or older;
2. Patient willing and able to provide a signed Patient Informed Consent Form;
3. Has a midline primary ventral, umbilical or incisional hernia;
4. Scheduled for a laparoscopic IPOM hernia repair;
5. Hernia can be successfully repaired with at least a 5 cm overlap of the mesh on all sides of the defect

Key Exclusion Criteria:

1. Patient has a known or suspected hypersensitivity to the constituent polymer of the investigational device, mesh, or other surgical products (e.g., sutures);
2. BMI > 40;
3. Patient is a current smoker, defined as self-reporting smoking more than 1 cigarette per day;
4. Patient is taking systemic immunosuppressive medications, systemic steroids, or chemotherapy at the time of informed consent;
5. Patient is pregnant, plans to become pregnant during the study period, or is breastfeeding;
6. Patient with Type 1 or uncontrolled Type 2 Diabetes Mellitus;
7. Patient has more than one hernia defect (to be confirmed intraoperatively);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2026-07-04 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Device Effect (SADEs) | through 12 months post-surgery
  Cumulative incidence of complications (CIC) related to the TAHRS including:
  Infection, Chronic pain, Recurrence of hernia, Impaired/delayed healing at the surgical site(s), Allergic reaction/hypersensitivity reaction,

SECONDARY OUTCOMES:
Rate of hernia recurrence through 12 months post- surgery | through 12 months post-surgery

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (4):
  - Ziekenhuis Oost-Limburg [ZOL], Genk, Limburg
  - Imelda Hospital, Bonheiden
  - AZ Sint-Jan, Ruddershove
  - CHU UCL Namur, Yvoir
- Universitary Hospital Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: No